CLINICAL TRIAL: NCT03720808
Title: The Comparison Of The Efficacy Of Three Methods Applied During Venous Blood Sampling On Reducing Pain And Fear In Children
Brief Title: Venous Blood Sampling-Related Pain and Fear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, İLKNUR GÖL, PhD RN, Asistant PROFESSOR, Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SY200217B06
Record Dates: First submitted 2018-10-24; First posted 2018-10-25 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Pain; Fear
Keywords: pain management; pain in children; venous blood sample; non-pharmacological method
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Balloon Blowing (Experimental): Venous blood sampling started as the children exhaled to blow up the balloon. Until the venous blood procedure ended, they continued to blow up the balloons.
  Interventions: Other: Balloon Blowing
- Ball Squeezing (Experimental): Before the venous blood collecting procedure, a soft ball was given to the right hands of the children and they were asked to squeeze and release this ball during the procedure.
  Interventions: Other: Ball Squeezing
- Coughing (Experimental): Just before the entrance of the needle, the child was asked to take a deep breath and the venous blood sampling procedure was started during coughing.
  Interventions: Other: Coughing
- Control (Experimental): No intervention was performed to reduce pain and fear in the control group.
  Interventions: Other: Control

INTERVENTIONS:
Other: Balloon Blowing — The parents of the children in this group were asked whether their children had the latex allergy or not and the children without the allergy were included in the group. The children's skills of blowing balloon were observed before the procedure. Before starting the venous blood sampling procedure, the children were asked to choose a balloon in the color they preferred and to start blowing the balloon at least 20 seconds before the procedure. Venous blood sampling started as the children exhaled to blow up the balloon. Until the venous blood procedure ended, they continued to blow up the balloons.
  Arms: Balloon Blowing
Other: Ball Squeezing — Before the venous blood collecting procedure, a soft ball was given to the right hands of the children and they were asked to squeeze and release this ball during the procedure.
  Arms: Ball Squeezing
Other: Coughing — The children included in this group were asked to cough after taking a deep breath during the venous blood sampling procedure. Before the procedure, the researcher showed the children how they should cough and asked them to imitate. The venous blood sampling was not performed until the child successfully completed coughing. The child was directed by the researcher during the procedure. Just before the entrance of the needle, the child was asked to take a deep breath and the venous blood sampling procedure was started during coughing.
  Arms: Coughing
Other: Control — No intervention was performed to reduce pain and fear in the control group.
  Arms: Control

SUMMARY:
This study is an experimental randomized controlled study conducted to compare the effect of balloon blowing, coughing, and ball squeezing methods applied during venous blood sampling from on pain and fear level in 7-12 year-old children. The population of the study consisted of all 7-12 year-old children who were referred to the blood-letting room for venous blood sampling in a state hospital. The sample of the study was determined as 120 children with confidence level of 95% and theoretical power of 95%. The children were divided into 4 groups of 30 people, including balloon blowing, ball squeezing, coughing, and control groups. Each intervention and control group was matched in terms of gender. In the study, the randomization of the sample group was performed by using stratification and block randomization methods.

DETAILED DESCRIPTION:
The study is a randomized controlled, non-blinded, experimental trial. The population of the study consisted of all 7-12 year-old children who came to the venipuncture room in the state hospital.It is stated in the literature that the sample size should be determined as minimum 30 in both experimental and control groups in the experimental studies and parametric measurements. Therefore, in the study, each group included 30 children including three experimental groups and a control group and in the power analysis, power of the study was found as 0.95 at the confidence level of 95%. In order to prevent bias and increase the validity of the data, the pain and fear scores of the children before and after the procedure were assessed by three different groups as children participating in the study (n:120), their parents as the people who know the children best (n:120), and a researcher specialized in pediatric nursing (n:1), and the inter-observer agreement was examined. The level of pain was assessed by the Wong Baker Faces Scale and the fear of pain was assessed by the Children's Fear Scale.

In this experimental study, the children and their parents who came to the venipuncture room for venous blood sampling were evaluated in terms of the inclusion criteria and the children and parents who did not meet the criteria were excluded from the study. The children and parents complying with the inclusion criteria were informed about the study and their written and verbal consents were received. The children were included in one of the 4 study groups, including the balloon blowing, coughing, ball squeezing, and the control group without any intervention. In the studies, it was determined that gender had an important effect on evaluation of pain.39,40 In order to control the effect of gender on pain, the children were stratified into study groups based on their gender and selected by using block randomization method in four study groups. The children were randomized to the related study group by drawing one of the study groups in the cloth bags prepared for the girls (pink) and the boys (blue). Papers with the same color and folding pattern representing the four groups (1,2,3,4) were thrown in the bags. In order to provide a randomized distribution and to reduce all negative effects, the children were asked to take randomly a paper from the bag according to the gender after making the necessary explanation to the parents and their children so that the groups became self-balancing. A total of 30 children including 15 girls and 15 boys were included in each group after intervention and control groups were matched in themselves in terms of gender. The study followed the CONSORT guideline for reporting randomized controlled trials.

ELIGIBILITY:
Inclusion Criteria:

The children,

* who were aged between 7-12 years,
* were healthy,
* did not receive any analgesic within the last 6 hours before venipuncture procedure,
* had no history of syncope during venipuncture procedure,
* agreed to participate in the study and gave the verbal and written consent.

Also, the parents were eligible for participation when meeting the following inclusion criteria:

* be healthy in terms of neurological functions,
* communicate verbally,
* understand and read Turkish,
* voluntarily sign the written informed consent.

Exclusion Criteria:

The children;

* who had neuro-developmental disorder,
* could not communicate verbally,
* had hearing and visual impairment,
* suffered from acute pyretic disease,
* received topical anesthesia, took any analgesic within the last 6 hours before venipuncture procedure,
* had chronic disease requiring frequent venipuncture.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Pain severity | 5 MONTHS
  The children and the parents were informed about the Wong Baker Faces Pain Rating Scale and they were asked to mark the children's pain levels on the scale 5 minutes before and after the venipuncture procedure. In addition, the pain levels of the children before and after the procedure were determined by the researcher who is a specialist in pediatric nursing by using the same scales.
  Wong Baker Faces Pain Rating Scale was developed by Donna Wong and Connie Morain Baker in 1981 and revised in 1983. The scale is one of the commonly used scales for measuring pain severity in children aged between 3-18 years. This scale has the faces and the pain score is determined according to the numerical values given to the faces. While smiley face "0 point" shows lack of pain, crying face "10 points" refer to severe pain.

SECONDARY OUTCOMES:
Fear levels | 5 MONTHS
  The children and the parents were informed about the Children's Fear Scale and they were asked to mark the children's fear levels on the scale within 5 mins before and after the venipuncture procedure. In addition, the fear levels of the children before and after the procedure were determined by the researcher who is a specialist in pediatric nursing by using the same scales.
  Children's Fear Scales has five facial expression and the fear is scored according to the numerical values given to the faces on the scale. The leftmost face "0 point" in the scale represents that the child has no fear and the rightmost face "4 points" represent that the child is frightened a lot.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu AYKANAT GİRGİN, PhD.RN, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Çankırı Karatekin Univesity, Çankiri, Turkey (Türkiye)